CLINICAL TRIAL: NCT04093440
Title: CardiOmetabolic SyndroME Response to Therapeutic lIfestyle Changes
Acronym: COSMETIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Holy Cross Hospital, Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCV-19-001
Record Dates: First submitted 2019-09-05; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Syndrome; ASCVD; Lifestyle Risk Reduction
Keywords: cardiometabolic clinic
MeSH Terms: conditions — Metabolic Syndrome; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation (Other): lifestyle modification: nutrition counselling, diet and physical exercise monitoring, smoking cessation, and medication optimization
  Interventions: Other: lifestyle modification

INTERVENTIONS:
Other: lifestyle modification — nutrition counselling, diet and physical exercise monitoring, smoking cessation, and medication optimization

SUMMARY:
Intensive lifestyle intervention has shown to be effective in high risk patient populations and has gathered support from leaders-as outlined in the 2015 consensus paper by the Cardiometabolic Health Alliance. Thus there has been a call to establish new care models that assist Metabolic Syndrome patients in reducing there risk. The investigators aim to evaluate the impact of a lifestyle intervention program on metabolic syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome patients meeting 3 of 5 criteria:

  1. waist circumference (37 in) in white and AA men, (35 in) in Asian men, and (31.5 in) in women;
  2. triglycerides ≥150 mg/dl;
  3. high-density lipoprotein cholesterol (HDL-C) <40 mg/dl in men and <50 mg/dl in women;
  4. blood pressure ≥130/85 mm Hg
  5. fasting glucose ≥100 mg/d or HgbA1c ≥ 5.71 (includes diabetics)
* Patients requiring secondary ASCD prevention

Exclusion Criteria:

* Patients with less than 5 year survival
* Patients with cancer undergoing therapy or on palliative treatment
* Patients with end stage heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Reversal of metabolic syndrome | At the end of 12 months
  Change in number of metabolic syndrome risk factors

SECONDARY OUTCOMES:
Mortality | within three to five years of intervention
  KM curve of patients with change in metabolic risk factors vs those with no change
hemoglobin A1c | At the end of 12 months
  change in hemoglobin A1c (percentage)
waist circumference | At the end of 12 months
  change in waist circumference (inches)
blood pressure | At the end of 12 months
  change in average blood pressure (mmHg)
total cholesterol | At the end of 12 months
  change in total cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Russo, MD, Principal Investigator — Jim Moran Heart and Vascular Research Center at Holy Cross Hospital; Paul Papagni, JD, Study Director — Jim Moran Heart and Vascular Research Center at Holy Cross Hospital
Locations (1):
- Internal Medicine Residency Clinic at Holy Cross Hospital, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No